CLINICAL TRIAL: NCT03577275
Title: A Randomised, Partially Double Blind, Placebo and Positive Controlled, 4 Way Crossover Study to Evaluate the Effect of Icosabutate (NST 4016) on the QT/QTc Interval in Healthy Subjects
Brief Title: A Study to Evaluate the Effects of NST-4016 on QT/Corrected QT (QTc) Interval
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NorthSea Therapeutics B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NST-01
Record Dates: First submitted 2018-06-22; First posted 2018-07-05 (Actual); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — icosabutate; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo oral capsule (Placebo Comparator): Single dose of placebo to match NST-4016
  Interventions: Drug: Placebo oral capsule
- Moxifloxacin 400mg (Active Comparator): Single 400mg dose of active comparator moxifloxacin (open label)
  Interventions: Drug: Moxifloxacin 400mg
- NST-4016 600mg (Experimental): Likely therapeutic dose of NST-4016
  Interventions: Drug: NST-4016 600mg
- NST-4016 2000mg (Experimental): Supratherapeutic dose of NST-4016
  Interventions: Drug: NST-4016 2000mg

INTERVENTIONS:
Drug: NST-4016 600mg — Likely maximum therapeutic dose of NST-4016
  Other Names: Icosabutate
  Arms: NST-4016 600mg
Drug: Placebo oral capsule — Placebo for comparison with moxifloxacin and potential NST-4016 effects
  Arms: Placebo oral capsule
Drug: Moxifloxacin 400mg — Active comparator with known effect on QT interval
  Arms: Moxifloxacin 400mg
Drug: NST-4016 2000mg — Supratherapeutic dose of NST-4016
  Other Names: Icosabutate
  Arms: NST-4016 2000mg

SUMMARY:
This is a Phase 1, single centre, randomised, double blind (except for moxifloxacin), placebo and positive controlled, 4 way crossover study assessing the ECG effects of therapeutic and supratherapeutic doses of icosabutate in healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males or females, of any race, between 18 and 55 years of age, inclusive, at Screening.
* 2. Body mass index (BMI) between 18.0 and 33.0 kg/m2, inclusive, at Screening
* 3. In good health

Exclusion Criteria:

* 1. An uninterpretable or abnormal ECG at Screening and/or Check in
* 2. History of risk factors for Torsades de Pointes
* 3. sustained supine systolic blood pressure >140 mmHg or <90 mmHg
* 4. Unstable cardiovascular disease, including recent myocardial infarction or cardiac arrhythmia.
* 5. Female subjects who are pregnant (or planning to become pregnant within 90 days after the final dose administration) or are currently lactating
* 6. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit (CRU) Ltd, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a cross over study so 32 subjects each completed 4 treatment arms
Groups:
- All Study Participants: This was a 4 way crossover study in which all study participants received the following treatments in random order; NST-4016 2000mg: Supratherapeutic dose of NST-4016, NST-4016 600mg: Likely maximum therapeutic dose of NST-4016, Moxifloxacin 400mg: Active comparator with known effect on QT interval, Placebo oral capsule: Placebo for comparison with moxifloxacin and potential NST-4016 effects. There were 12 possible treatment sequences
Period: Overall Study
Arm/Group | All Study Participants
Started | 32 (All participants received all of the 4 interventions)
Placebo | 32
Moxifloxacin 400mg | 32
NST-4016 600mg | 32
NST-4016 2000mg | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants were randomized to receive all 4 interventions
Arm/Group | All Study Participants
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 24
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 32

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fridericia's Correction for QT Interval (QTcF)
Description: Electrocardiogram measurement of the maximum absolute change from baseline in Fridericia's correction for QT interval (QTcF)
Time Frame: 24 hours
Population: The primary endpoint for this trial was the placebo corrected change from baseline in QTcF. The data presented here are the maximum absolute change from baseline for placebo, moxifloxacin 400mg, NST-4016 600mg and NST-4016 2000mg.
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Placebo Oral Capsule | Moxifloxacin 400mg | NST-4016 600mg | NST-4016 2000mg
Number analyzed (Participants) | 32 | 32 | 32 | 32
msec | -4.6 (1.52) | 11.5 (0.88) | -6.0 (1.39) | -6.1 (1.42)
Statistical Analysis 1: Comparison: Placebo Oral Capsule vs Moxifloxacin 400mg vs NST-4016 600mg vs NST-4016 2000mg; The primary analysis was based on concentration-QTc modeling of the relationship between icosabutate and delta delta QTcF, with the intent to exclude an effect > 10 msec at clinically relevant icosabutate plasma concentrations. Assay sensitivity was evaluated by concentration-QTc analysis of the effect on delta delta QTcF of moxifloxacin using a similar model as for the primary analysis; Test type: Other; The primary analysis was based on concentration-QTc modeling of the relationship between icosabutate and delta delta QTcF, with the intent to exclude an effect > 10 msec at clinically relevant icosabutate plasma concentrations

2. Secondary Outcome: Change From Baseline in Heart Rate (HR)
Description: Electrocardiogram measurement of change from baseline in heart rate (HR) maximum values presented
Time Frame: 24 hours
Population: maximum values of change in heart rate from baseline over the 24 hours post dose
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Groups:
- Placebo: Single dose of placebo to match NST-4016 Placebo oral capsule: Placebo for comparison with moxifloxacin and potential NST-4016 effects
- Moxifloxacin 400mg: Single 400mg dose of active comparator moxifloxacin (open label) Moxifloxacin 400mg: Active comparator with known effect on QT interval
- NST-4016 600mg: Likely therapeutic dose of NST-4016 NST-4016 600mg: Likely maximum therapeutic dose of NST-4016
- NST-4016 2000mg: Supratherapeutic dose of NST-4016 NST-4016 2000mg: Supratherapeutic dose of NST-4016
Arm/Group | Placebo | Moxifloxacin 400mg | NST-4016 600mg | NST-4016 2000mg
Number analyzed (Participants) | 32 | 32 | 32 | 32
beats per minute | 9.9 (0.86) | 12.2 (0.85) | 12.6 (0.88) | 15.6 (0.85)

3. Secondary Outcome: Change From Baseline in Fridericia's Correction for QT Interval (QTcF)
Description: Electrocardiogram measurement of change from baseline in Fridericia's correction for QT interval (QTcF)
Time Frame: 24 hours
Population: The largest change in QTcF for each arm during the study is presented below
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Placebo | Moxifloxacin 400mg | NST-4016 600mg | NST-4016 2000mg
Number analyzed (Participants) | 32 | 32 | 32 | 32
msec | -4.6 (1.52) | 11.5 (0.88) | -6.0 (1.39) | -5.7 (1.39)

4. Secondary Outcome: Change From Baseline in PR Interval (PR)
Description: Electrocardiogram measurement of change from baseline in PR interval (PR)
Time Frame: 24 hours
Population: maximum change from baseline during the study period is reported
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Placebo | Moxifloxacin 400mg | NST-4016 600mg | NST-4016 2000mg
Number analyzed (Participants) | 32 | 32 | 32 | 32
msec | -11.0 (1.32) | -11.9 (1.30) | -11.4 (1.36) | -12.4 (1.30)

5. Secondary Outcome: Change From Baseline in QRS Interval (QRS)
Description: Electrocardiogram measurement of change from baseline in QRS interval (QRS)
Time Frame: 2 hours
Population: The data presented is from the 2 hour time point corresponding to T max
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Placebo | Moxifloxacin 400mg | NST-4016 600mg | NST-4016 2000mg
Number analyzed (Participants) | 32 | 32 | 32 | 32
msec | -0.2 (0.17) | -0.1 (0.16) | -0.2 (0.17) | 0.2 (0.16)

ADVERSE EVENTS:
Time Frame: 3.5 months
Arm/Group | Placebo Oral Capsule | Moxifloxacin 400mg | NST-4016 600mg | NST-4016 2000mg
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 1/32
Other Adverse Events (participants affected / at risk) | 4/32 | 6/32 | 4/32 | 15/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Oral Capsule (N=32) | Moxifloxacin 400mg (N=32) | NST-4016 600mg (N=32) | NST-4016 2000mg (N=32)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — One subject (female) experienced an SAE of cerebrovascular accident that began <17 days post the last dose of the study drug (600 mg icosabutate in Dosing Period 4). The Investigator considered the event to be severe and related to the study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Oral Capsule (N=32) | Moxifloxacin 400mg (N=32) | NST-4016 600mg (N=32) | NST-4016 2000mg (N=32)
Gastrointestinal disturbance (Gastrointestinal disorders) | 4 (4) | 6 (6) | 4 (4) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT03577275/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT03577275/SAP_001.pdf